CLINICAL TRIAL: NCT03152773
Title: Heart Catheterization Using Magnetic Resonance Imaging (MRI) Fluoroscopy and Passive Guidewires
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The enrollment has been on hold since 2022 because the MRI scanner aging has made it inadequate for human catheter procedures.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 170095; 17-H-0095
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01-20

CONDITIONS: Pulmonary Artery Hypertension; Congenital Heart Disease; Structural Heart Disease
Keywords: MRI Catheterization; Real-time MRI
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Heart Defects, Congenital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Open label
  Interventions: Procedure: MRI Heart guidewire catheterization

INTERVENTIONS:
Procedure: MRI Heart guidewire catheterization — to conduct left and right heart guidewire catheterization using real-time MRI fluoroscopy in human research subjects already undergoing medically necessary left and right heart catheterization. We will use only passive MRI-compatible catheters and a specific guidewire shown to be safe under specific conditions. Under the conditions of use, the guidewire is not susceptible to heating.

SUMMARY:
Background:

A heart catheterization is a diagnostic heart procedure used to measure pressures and take pictures of the blood flow through the heart chambers. Magnetic resonance imaging (MRI) fluoroscopy shows continuous pictures of the heart chambers that doctors can watch while they work. Researchers want to test this procedure with catheterization tools routinely used in x-ray catheterization called guidewires. Guidewires will help move the heart catheter through the different heart chambers. Guidewires are usually considered unsafe during MRI because MRI can cause a guidewire to heat while inside the blood vessels and heart. Researchers are testing special low energy MRI settings that allow certain guidewires to be used during MRI catheterization without heating. Using these guidewires during MRI may help to decrease the amount of time you are in the MRI scanner, and the overall time the MRI catheterization procedure takes.

Objectives:

To test if certain MRI settings make it safe to use a guidewire during MRI fluoroscopy.

Eligibility:

Adults 18 and older whose doctors have recommended right heart catheterization.

Design:

Researchers will screen participants by reviewing their lab results and questionnaire answers.

Participants may give 4 blood samples.

Participants will be sedated. They will have a tube (catheter) placed in the groin, arm, or neck if they don t already have one.

Patches on the skin will monitor heart rhythm. Special antennas, covered in pads, will be placed against the body.

Participants will lie flat on a table that slides in and out of the MRI scanner as it makes pictures. Participants will get earplugs for the loud knocking noise. They can talk on an intercom. They will be inside the scanner for up to 2 hours. They can ask to stop at any time.

During a heart catheterization, catheters will be inserted through the tubes already in place. The catheters are guided by MRI fluoroscopy into the chambers of the heart and vessels. The guidewire will help position the catheter.

DETAILED DESCRIPTION:
Heart catheterization is a minimally invasive procedure to measure pressure into specific heart cavities. Heart catheterization usually uses X-ray guidance, which involves radiation exposure, and which fails to visualize soft tissue. For several years, real-time magnetic resonance imaging (MRI) fluoroscopy has been the standard technique to guide right heart catheterization at the NIH clinical center.

Guidewires are standard tools used to steer catheters through the body and heart. Guidewires have not been used during MRI fluoroscopy catheterization because of the risk of heating. We have developed MRI techniques that do not risk heating using specific commercial guidewires. In this protocol we will use this new low-energy real-time MRI fluoroscopy technique to enable use of guidewires during otherwise standard MRI catheterization of the right side of the heart through veins, and of the left side of the heart through the aorta.

In the second phase of the protocol, we will begin performing systematic MRI guidewire heart catheterization without X-ray whenever possible. We will assess the heart s response to hemodynamic provocation during MRI catheterization tailored to the patient s problem. We will use this protocol to further refine the technique.

This will enable future testing of devices for adult and pediatric MRI-fluoroscopy catheterization, which may lead to new non-surgical treatments of cardiovascular disease.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 years old
* Undergoing medically necessary diagnostic or interventional right cardiovascular catheterization, alone or in combination with a left cardiovascular catheterization

EXCLUSION CRITERIA:

* Cardiovascular instability including ongoing acute myocardial infarction, refractory angina or ischemia, and decompensated congestive heart failure.
* Women who are pregnant or nursing
* Unable to undergo magnetic resonance imaging

  * Cerebral aneurysm clip
  * Neural stimulator (e.g. TENS-Unit)
  * Any type of ear implant
  * Ocular foreign body (e.g. metal shavings)
  * Metal shrapnel or bullet.
  * Any implanted device (e.g. insulin pump, drug infusion device), unless it is labeled safe for MRI

EXCLUSION CRITERIA FOR GADOLINIUM-BASED CONTRAST AGENTS:

Renal excretory dysfunction, estimated glomerular filtration rate < 30 mL/min/1.73m2 body surface area according to the Modification of Diet in Renal Disease criteria

Glomerular filtration rate will be estimated using the CKD-EPI equation:

eGFR = 141 x (minimum of (S(Cr)/k, 1)^alpha x (maximum of (S(Cr) /k, 1))^-1.209 x 0.993^Age x 1.018 (if female) x 1.159 (if black)

Where

S(Cr) = serum creatinine

alpha = -0.329 for females and -0.411 for males

k = 0.7 for females and 0.9 for males

Subjects meeting this exclusion criterion may still be included in the study but may not be exposed to gadolinium-based contrast agents.

Exclusion criteria for ferumoxytol:

* Allergy to ferumoxytol or to mannitol excipient
* Does not wish to be exposed to ferumoxytol

Exclusion criteria for MRI left heart catheterization:

-Severe aortic valve stenosis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
The principal objective of this protocol is to test the safety and feasibility of MRI fluoroscopy catheter navigation using 0.035 guidewires during left and right heart catheterization guided by low-SAR MRI pulse sequences | 2 hours
  Acquisition of hemodynamic and saturation data from targeted chambers and vessels.

SECONDARY OUTCOMES:
Additional objectives are to test and enhanced MRI as an adjunct to routine hemodynamic cardiac catheterization | 2 hours
  Conspicuity of Glidewires during MRI fluoroscopy catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Lederman, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The authors are willing to share de-identified subject data upon reasonable request

REFERENCES:
- [Derived] Campbell-Washburn AE, Rogers T, Stine AM, Khan JM, Ramasawmy R, Schenke WH, McGuirt DR, Mazal JR, Grant LP, Grant EK, Herzka DA, Lederman RJ. Right heart catheterization using metallic guidewires and low SAR cardiovascular magnetic resonance fluoroscopy at 1.5 Tesla: first in human experience. J Cardiovasc Magn Reson. 2018 Jun 21;20(1):41. doi: 10.1186/s12968-018-0458-7. PMID 29925397
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-H-0095.html